CLINICAL TRIAL: NCT06054269
Title: Randomized Controlled Trial, Double Blind, Phase III, to Evaluate the Immunogenicity of an Adjuvanted Influenza Vaccine Among Health Care Personnel (EDUCATE)
Brief Title: Clinical Trial to Evaluate the Immunogenicity of an Adjuvanted Influenza Vaccine Among HCP
Acronym: EDUCATE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Peruvian Clinical Research (Other); Hospital Nacional Cayetano Heredia (Unknown); Hospital Nacional Arzobispo Loayza (Other); U.S. Naval Medical Research Unit No.6 (NAMRU-6) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NAMRU6.2019.0011
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FLUAD Quadrivalent (Experimental): Participants administered a single dose of adjuvanted egg-based quadrivalent influenza vaccine (FLUAD Quadrivalent by Seqirus, 15 µg of HA from each strain).
  Interventions: Biological: FLUAD Quadrivalent
- FluQuadri (Active Comparator): Participants administered a single dose of standard dose egg-based quadrivalent influenza vaccine (FluQuadri by Sanofi-Pasteur, 15 µg of HA from each strain).
  Interventions: Biological: FluQuadri

INTERVENTIONS:
Biological: FLUAD Quadrivalent — 0.5 mL intramuscular dose of FLUAD Quadrivalent
  Arms: FLUAD Quadrivalent
Biological: FluQuadri — 0.5 mL intramuscular dose of FluQuadri
  Arms: FluQuadri

SUMMARY:
This randomized, double-blinded trial will assess humoral immune responses to adjuvanted, egg-based quadrivalent influenza vaccines compared to standard dose, egg-based quadrivalent influenza vaccines among healthcare personnel (HCP). The trial will be conducted at two sites in Lima, Peru during 2022 and 2023.

DETAILED DESCRIPTION:
The trial will be conducted at two hospital sites in Lima, Peru during 2022-2023 among HCP who were previously enrolled in the Cohort study of Influenza and other Respiratory Viruses among HCP in Peru (cohort size: approximately 1500 participants). The minimum number of participants to be enrolled is 248 in total (142 subjects per vaccine group), and the aim is to enroll approximately 800 participants (400 subjects per vaccine group). The study design is a randomized, double-blind vaccine trial. Eligible HCP at each site who consent to participate will be randomized 1:1 to receive either a single dose of adjuvanted egg-based quadrivalent influenza vaccine (AD, FLUAD Quadrivalent by Seqirus, 15 µg of hemagglutinin [HA] from each strain) or standard dose, egg-based quadrivalent influenza vaccine (SD, FluQuadri by Sanofi-Pasteur, 15 µg of HA from each strain).

Participants will be invited to come to the study site to be screened for eligibility to participate in the clinical trial. After they consent to participate and sign informed consent form, participants will visit the site for medical assessment and vaccination. Additional brief medical adverse event assessments will be performed on days 3 and 7. Participants will be followed up to twice per week via SMS or phone calls to assess if they become sick with a respiratory event. In the event they become sick, they will be asked questions about their illness through an acute illness survey and a mid-turbinate nasal swab specimen will be collected and tested for influenza virus. Additional surveys will be administered on day 28 post-vaccination as well as at the end of the influenza season.

Participants will have blood collected just prior to vaccination (Day 0) and at approximately 28 days and 6 months post-vaccination (or at the end of influenza virus circulation as determined by active surveillance data) to evaluate humoral immune responses to vaccination. After these specimens are tested, differences in seroconversion and seroprotection between AD and SD vaccination groups will be assessed. In addition, we multivariable modelling will be used to assess risk factors for poor immunogenicity and to assess possible effects of repeated vaccination.

As an optional sub-study, indicators of cell-mediated immune (CMI) responses to influenza vaccination will be examined. This part of the study, which is optional to participants, will require collection of additional blood samples at prior to vaccination (Day 0) and at 7 and 28 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Have participated in the healthcare personnel cohort study at Hospital Nacional Cayetano Heredia or Hospital Nacional Arzobispo Loayza during 2016-2021;
* Work at the facility full-time (≥30 hours per week);
* Have routine, direct, hands-on or face-to-face contact with patients (≤1 meter) as part of a typical work shift, including, but not limited to, physicians, nurses, respiratory therapists, physical therapists, unit clerks, radiograph technicians, medical assistants, and transporters;
* Work at the facility for ≥1 year prior to enrollment and planning to continue working at the facility for one year after enrollment;
* Willing to receive influenza vaccination (adjuvanted or standard dose);
* Women of childbearing age must complete the following criteria to be eligible:

  1. Have a negative urine pregnancy test performed by the study staff ≤24 hours preceding receipt of the vaccine;
  2. Be willing to use a reliable form of contraception approved by the Investigator for ≤2 months after receiving the vaccine. If they are not currently using an approved contraceptive, study staff will provide access to contraceptives;
  3. Must not be breastfeeding.

Exclusion Criteria:

* Have received a vaccine against influenza during the 2022 influenza season (season of clinical trial);
* Have a severe, life-threatening allergy to influenza vaccines, eggs, or influenza vaccine components;
* Have a history of Guillain-Barre Syndrome or other autoimmune diseases;
* Received blood or blood products within 3 months of enrollment;
* Be pregnant, confirmed by rapid pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Soto, MD, MPH, Principal Investigator — Naval Medical Research Unit- 6; Roger Antonio Hernandez Diaz, MD, MSc, Principal Investigator — Hospital Nacional Cayetano Heredia; Eduardo Demetrio Matos Prado, MD, Principal Investigator — Hospital Nacional Arzobispo Loayza
Locations (2):
- Peru (2):
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Cayetano Heredia, Lima

IPD SHARING:
Plan to Share IPD: No
No current plans to share IPD

REFERENCES:
- [Derived] Marcenac P, Soto G, Yau T, Carreon JD, Romero C, Gonzales M, La Rosa S, Arriola CS, Prouty M, Diaz RAH, Romero FA, Llanos-Cuentas A, Prado EDM, Silva M, Fowlkes A, Levine MZ, Azziz-Baumgartner E, Duca LM, Neyra J. Comparison of the immunogenicity of adjuvanted and conventional egg-based quadrivalent influenza vaccines among healthcare personnel in Lima, Peru: A randomized controlled trial. Int J Infect Dis. 2026 Jan;162:108205. doi: 10.1016/j.ijid.2025.108205. Epub 2025 Nov 11. PMID 41232749

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLUAD Quadrivalent | FluQuadri
Started | 95 | 97
Provided 28 Days Post-vaccination Blood Specimen | 95 | 95
Provided 6 Months Post-vaccination Blood Specimen | 94 | 96
Completed | 95 | 97
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLUAD Quadrivalent | FluQuadri | Total
Number analyzed (Participants) | 95 | 97 | 192
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-50 years old | 47 | 56 | 103
  Age group: 50-65 years old | 46 | 34 | 80
  Age group: >65 years old | 2 | 7 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 39 | 41 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Mixed | 77 | 89 | 166
  Race/ethnicity: Quechua | 7 | 6 | 13
  Race/ethnicity: African Peruvian | 4 | 2 | 6
  Race/ethnicity: Caucasian | 3 | 0 | 3
  Race/ethnicity: Asian | 2 | 0 | 2
  Race/ethnicity: Aymara | 2 | 0 | 2
Body mass index [Count of Participants; unit: Participants]
  Healthy (18.5-24.9) | 10 | 16 | 26
  Overweight (25.0-29.9) | 50 | 45 | 95
  Obese (>=30.0) | 35 | 36 | 71
Current smoking habit [Count of Participants; unit: Participants]
  Non-smoker | 85 | 91 | 176
  Smoke periodically-daily | 10 | 6 | 16
History of chronic conditions [Count of Participants; unit: Participants]
  No | 81 | 81 | 162
  Yes | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Geometric Mean Titers (GMT) Post-vaccination (Day 28) of Each Vaccine Reference Virus
Description: The geometric mean of antibody titers after a single dose of FLUAD Quadrivalent (adjuvanted dose, AD) vs. FluQuadri (standard dose, SD) as measured by HI assay for egg-grown influenza A(H1N1)pdm09, A(H3N2), B/Yamagata, and B/Victoria vaccine reference viruses at approximately 28 days post-vaccination
Time Frame: 28 days post-vaccination
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: antibody titer
Arm/Group | FLUAD Quadrivalent | FluQuadri
Number analyzed (Participants) | 95 | 95
antibody titer
  Influenza A(H1N1)pdm09 | 584.2 [453.1 to 753.3] | 342.8 [265.9 to 442.0]
  Influenza A(H3N2) | 217.4 [173.0 to 273.1] | 169.0 [134.5 to 212.3]
  Influenza B/Victoria | 102.1 [76.5 to 136.2] | 107.8 [80.8 to 143.9]
  Influenza B/Yamagata | 211.1 [170.5 to 261.4] | 184.4 [148.9 to 228.4]
Statistical Analysis 1: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination geometric mean antibody titers to the influenza A(H1N1)pdm09 vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination geometric mean antibody titers to the influenza A(H3N2) vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.066, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination geometric mean antibody titers to the influenza B/Victoria vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.694, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination geometric mean antibody titers to the influenza B/Yamagata vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.408, Wilcoxon (Mann-Whitney)

2. Primary Outcome: HI GMT Post-vaccination (6 Months) of Each Vaccine Reference Virus
Description: The geometric mean of antibody titers after a single dose of AD vs SD vaccine as measured by HI assay for egg-grown influenza A(H1N1)pdm09, A(H3N2), B/Yamagata, and B/Victoria vaccine reference viruses at approximately 6 months post-vaccination
Time Frame: 6 months post-vaccination
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: antibody titer
Arm/Group | FLUAD Quadrivalent | FluQuadri
Number analyzed (Participants) | 94 | 96
antibody titer
  Influenza A(H1N1)pdm09 | 177.4 [137.2 to 229.3] | 128.4 [99.6 to 165.5]
  Influenza A(H3N2) | 94.1 [75.0 to 118.0] | 67.2 [53.7 to 84.1]
  Influenza B/Victoria | 34.5 [25.8 to 46.1] | 41.2 [30.9 to 54.9]
  Influenza B/Yamagata | 55.5 [43.2 to 71.4] | 57.0 [44.4 to 73.0]
Statistical Analysis 1: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.164, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.113, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.404, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.879, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Seroconversion Rate (SCR) to Each Vaccine Reference Virus Post-vaccination
Description: The percent of participants with paired samples that achieved ≥4-fold rises comparing post- (approximately 28 days) versus pre-vaccination titers, and post-vaccination titers ≥40 for each vaccine reference virus (egg-grown influenza A(H1N1)pdm09, A(H3N2), B/Yamagata, and B/Victoria vaccine reference viruses) following a single dose of AD vs. SD vaccine.
Time Frame: 28 days post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FLUAD Quadrivalent | FluQuadri
Number analyzed (Participants) | 95 | 95
percentage of participants
  Influenza A(H1N1)pdm09 | 88.4 [80.4 to 93.4] | 62.1 [52.1 to 71.2]
  Influenza A(H3N2) | 82.1 [73.2 to 88.5] | 62.1 [52.1 to 71.2]
  Influenza B/Victoria | 47.4 [37.6 to 57.3] | 52.6 [42.7 to 62.4]
  Influenza B/Yamagata | 63.2 [53.1 to 72.2] | 49.5 [39.6 to 59.4]
Statistical Analysis 1: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroconversion rate to the influenza A(H1N1)pdm09 vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroconversion rate to the influenza A(H3N2) vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.002, Chi-squared
Statistical Analysis 3: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroconversion rate to the influenza B/Victoria vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.468, Chi-squared
Statistical Analysis 4: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroconversion rate to the influenza B/Yamagata vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.057, Chi-squared

4. Primary Outcome: SCR to Each Vaccine Reference Virus Post-vaccination
Description: The percent of participants with paired samples that achieved ≥4-fold rises comparing post- (approximately 6 months) versus pre-vaccination titers, and post-vaccination titers ≥40 for each vaccine reference virus (egg-grown influenza A(H1N1)pdm09, A(H3N2), B/Yamagata, and B/Victoria vaccine reference viruses) following a single dose of AD vs. SD vaccine.
Time Frame: 6 months post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FLUAD Quadrivalent | FluQuadri
Number analyzed (Participants) | 94 | 96
percentage of participants
  Influenza A(H1N1)pdm09 | 53.2 [43.2 to 63.0] | 41.7 [32.3 to 51.7]
  Influenza A(H3N2) | 50.0 [40.1 to 59.9] | 39.6 [30.4 to 49.6]
  Influenza B/Victoria | 18.1 [11.6 to 27.1] | 28.1 [20.1 to 37.8]
  Influenza B/Yamagata | 16.0 [9.9 to 24.7] | 10.4 [5.8 to 18.1]
Statistical Analysis 1: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.112, Chi-squared
Statistical Analysis 2: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.149, Chi-squared
Statistical Analysis 3: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.101, Chi-squared
Statistical Analysis 4: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.259, Chi-squared

5. Primary Outcome: Seroprotection Rate (SPR) to Each Vaccine Reference Virus Post-vaccination
Description: The percent of participants with post-vaccination titers ≥40 for each vaccine reference virus (egg-grown influenza A(H1N1)pdm09, A(H3N2), B/Yamagata, and B/Victoria vaccine reference viruses) following a single dose of AD vs. SD vaccine.
Time Frame: 28 days post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FLUAD Quadrivalent | FluQuadri
Number analyzed (Participants) | 95 | 95
percentage of participants
  Influenza A(H1N1)pdm09 | 98.9 [94.3 to 99.9] | 94.7 [88.3 to 97.7]
  Influenza A(H3N2) | 95.8 [89.7 to 98.4] | 94.7 [88.3 to 97.7]
  Influenza B/Victoria | 81.1 [72.0 to 87.7] | 76.8 [67.4 to 84.2]
  Influenza B/Yamagata | 98.9 [94.3 to 99.9] | 96.8 [91.1 to 98.9]
Statistical Analysis 1: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroprotection rate to the influenza A(H1N1)pdm09 vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.097, Chi-squared
Statistical Analysis 2: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroprotection rate to the influenza A(H3N2) vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.733, Chi-squared
Statistical Analysis 3: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroprotection rate to the influenza B/Victoria vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.477, Chi-squared
Statistical Analysis 4: Comparison: FLUAD Quadrivalent vs FluQuadri; For comparison of post-vaccination seroprotection rate to the influenza B/Yamagata vaccine virus between recipients of FLUAD Quadrivalent and FluQuadri; Test type: Superiority; p = 0.312, Chi-squared

6. Primary Outcome: SPR to Each Vaccine Reference Virus Post-vaccination
Description: as for outcome 5
Time Frame: 6 months post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FLUAD Quadrivalent | FluQuadri
Number analyzed (Participants) | 94 | 96
percentage of participants
  Influenza A(H1N1)pdm09 | 93.6 [86.8 to 97.0] | 88.5 [80.6 to 93.5]
  Influenza A(H3N2) | 90.4 [82.8 to 94.9] | 74.0 [64.4 to 81.7]
  Influenza B/Victoria | 55.3 [45.3 to 65.0] | 56.2 [46.3 to 65.7]
  Influenza B/Yamagata | 73.4 [63.7 to 81.3] | 74.0 [64.4 to 81.7]
Statistical Analysis 1: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.220, Chi-squared
Statistical Analysis 2: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.003, Chi-squared
Statistical Analysis 3: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.897, Chi-squared
Statistical Analysis 4: Comparison: FLUAD Quadrivalent vs FluQuadri; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.931, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the moment of vaccination to the 7 days following vaccination. In the study, this corresponded to monitoring study participants from first enrollments in November 2022 to final enrollments in January 2023.
Arm/Group | FLUAD Quadrivalent | FluQuadri
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/97
Other Adverse Events (participants affected / at risk) | 70/95 | 61/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLUAD Quadrivalent (N=95) | FluQuadri (N=97)
Local pain at the vaccine injection site (Skin and subcutaneous tissue disorders) | 42 | 32
Headache (General disorders) | 14 | 16
Muscle/articular pain (Musculoskeletal and connective tissue disorders) | 15 | 7
Malaise (General disorders) | 12 | 5
Local swelling at the vaccine injection site (Skin and subcutaneous tissue disorders) | 7 | 4
Local induration at the vaccine injection site (Skin and subcutaneous tissue disorders) | 9 | 1
Local redness at the vaccine injection site (Skin and subcutaneous tissue disorders) | 5 | 3
Local itchiness at the vaccine injection site (Skin and subcutaneous tissue disorders) | 5 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Measured or subjective fever (General disorders) | 4 | 1
Nausea (General disorders) | 2 | 2
Lack of appetite (General disorders) | 1 | 2
Dizziness (General disorders) | 2 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Loose stool (Gastrointestinal disorders) | 0 | 2
Hematoma at the vaccine injection site (Skin and subcutaneous tissue disorders) | 1 | 2
Itchiness (Skin and subcutaneous tissue disorders) | 0 | 2
Increase of systolic blood pressure (Vascular disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Pain in left eye (Eye disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Right malar hematoma (Skin and subcutaneous tissue disorders) | 1 | 0
Hyposmia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Itchiness and rash (Skin and subcutaneous tissue disorders) | 0 | 1
Itchiness and rash at vaccine injection site (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT06054269/Prot_SAP_000.pdf